CLINICAL TRIAL: NCT03802552
Title: Comparative Pharmacokinetics and Pharmacodynamics (PK/PD) of Cefadroxil and Cephalexin for Pediatric Musculoskeletal (MSK) Infections
Brief Title: Cefadroxil and Cephalexin Drug Levels and Dosing in Pediatric Musculoskeletal Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-2142
Record Dates: First submitted 2018-12-26; First posted 2019-01-14 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Osteomyelitis; Septic Arthritis; Pyomyositis
MeSH Terms: conditions — Osteomyelitis; Arthritis, Infectious; Pyomyositis | interventions — Cefadroxil; Cephalexin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefadroxil then Cephalexin (Experimental): Receive cefadroxil first, then receive cephalexin after washout.
  Interventions: Drug: Cefadroxil; Drug: Cephalexin
- Cephalexin then Cefadroxil (Experimental): Receive cephalexin first, then receive cefadroxil after washout.
  Interventions: Drug: Cefadroxil; Drug: Cephalexin

INTERVENTIONS:
Drug: Cefadroxil — oral one-time dose of cefadroxil
  Other Names: Duricef
Drug: Cephalexin — oral one-time dose of cephalexin
  Other Names: Keflex

SUMMARY:
The goal of this study is to figure out the best doses for two antibiotics (called cefadroxil and cephalexin) when they are used to treat bone, joint, or muscle infections in children. In order to do this, the study will collect data about children admitted to Children's Hospital Colorado who have these types of infections. During the study, these patients will receive doses by mouth of each of these antibiotics, in addition to an IV antibiotic (given through a vein) used to treat their infection. After the dose of the first antibiotic, blood samples will be drawn every few hours to measure how much of the drug is still in their body, until it is all gone. After the first antibiotic is out of the patient's body, the same will be done for the second antibiotic. Measurements, in the lab, of how much of these antibiotics are needed to kill the most common bacteria causing these infections, which is a type of "Staph" bacteria called "MSSA", will be taken. Finally, the blood levels of the antibiotics and the information from the lab tests about the Staph bacteria will be used to calculate how much and how often of the antibiotic should be given to children with bone, joint, or muscle infections. Currently, these types of infections are treated with an antibiotic that children have to take four times every day. The goal of this study is to find an antibiotic that children can take only two or three times per day.

DETAILED DESCRIPTION:
This study aims to shift the current treatment paradigm for the use of oral first-generation cephalosporins in pediatric musculoskeletal (MSK) infections. Optimizing treatment for MSK infections is particularly important, as osteomyelitis is one of the most common severe infections affecting children. Treatment for these infections has markedly improved over the last few decades, but significant morbidity is still seen, including the possibility of permanent disability due to pathologic fracture, growth arrest, and joint destruction. To avoid these long term sequelae and recrudescent infection, early diagnosis, appropriate therapy, and prolonged treatment courses (typically 4-6 weeks, or longer) are essential.

The most commonly used antibiotic for MSK infections is cephalexin, a first-generation cephalosporin. It is well tolerated, provides good tissue penetration, and has a preferred spectrum of activity for typical MSK pathogens, including methicillin susceptible Staphylococcus aureus (MSSA). Despite cephalexin's widespread use, its most significant disadvantage is its short plasma half-life. Because of this, cephalexin is traditionally dosed four times daily (QID) for serious infections like osteomyelitis. However, this dosing frequency, especially for prolonged treatment courses, proves difficult for both patients and their families. Concern about poor adherence drives some providers to prolong IV therapy or dose cephalexin three times daily (TID), though there are insufficient pharmacokinetic/pharmacodynamic (PK/PD) or outcome data to support TID dosing.

Cefadroxil, another first-generation cephalosporin, is an appealing alternative to cephalexin due to its longer half-life. Because of this, the investigators hypothesize that cefadroxil could be used effectively in pediatric patients with MSK infections with a more convenient dosing schedule than cephalexin. While cephalexin is typically dosed 3-4 times per day, cefadroxil could likely be dosed 2-3 times per day, even for serious infections like osteomyelitis. However, cefadroxil is rarely prescribed to children due to a lack of pediatric PK/PD data to guide dosing. Our study aims to address this unmet need and help physicians use these existing drugs in smarter and more effective ways in pediatric MSK infections.

The specific aims of this study are to:

1. Use a Population PK approach to define comparative PK parameters of cefadroxil and cephalexin in pediatric patients with MSK infections (osteomyelitis, septic arthritis, pyomyositis).
2. Establish reference MIC ranges for both cefadroxil and cephalexin against MSSA isolates.
3. Perform pharmacodynamic modeling (Monte Carlo simulation) based on the above PK parameters and MIC data to evaluate the expected PK/PD target attainment of cefadroxil and cephalexin at different dosing intervals: cephalexin given as 3 vs. 4 divided doses per day; cefadroxil given as 2 vs. 3 doses against a range of MICs.

To answer these questions, patients with MSK infections admitted to Children's Hospital Colorado (CHCO) will be enrolled in this study and sequentially given doses of both cefadroxil and cephalexin. After each oral dose, serum levels of the antibiotic will be measured at set time points until the drug is expected to be fully cleared. They will then receive the second antibiotic after a 24-hour washout period. MIC ranges will be measured based on banked MSSA isolates. Based on these study-derived PK and MIC data, adequacy of the studied cephalexin and cefadroxil dosing regimens will be analyzed.

If the study is able to confirm a favorable PK/PD profile for twice daily (BID) and/or three times daily (TID) cefadroxil dosing in children, even for severe infections, it could have an immediate impact on prescribing habits. Less frequent dosing would be an improvement over the current standard of care, allowing for easier medication administration, improved adherence, and increased provider confidence for early transition to oral therapy, which are all essential for optimal treatment of pediatric MSK infections.

ELIGIBILITY:
Inclusion Criteria:

Children who are admitted to Children's Hospital Colorado and:

* Are to be treated for a deep musculoskeletal infection (osteomyelitis, septic arthritis, pyomyositis), as determined by their primary medical team
* Are aged 6 months to 18 years

Exclusion Criteria:

Patients will be excluded if they:

* Are less than 6 months of age or greater than 18 years of age
* Weigh less than 5.5 kg
* Weigh greater than the 95%ile for age
* Have underlying current renal disease based on medical history
* Have an underlying chronic medical condition-examples include cystic fibrosis, sickle cell anemia, inflammatory bowel disease, pancreatitis, hepatitis, immunodeficiency, cancer, spina bifida, chromosomal abnormalities, cerebral palsy, or metabolic disorders.
* Have a history of significant drug allergy to any beta-lactam antibiotic (e.g. anaphylaxis and/or angioedema)
* Are on an oral cephalosporin at time of enrollment
* Are started on an oral cephalosporin during the study

  o Note: If an enrolled patient is started on an oral cephalosporin prior to completion of the study, they will be removed from the study. However, data obtained prior to their receipt of an oral cephalosporin will still be included in the analysis.
* Are known to be pregnant

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Time above Minimum Inhibitory Concentration (T > MIC) | up to 24 hours
  As a surrogate of treatment efficacy for cefadroxil and cephalexin, the investigators will measure the time that free serum concentrations (T > MIC) of cefadroxil and cephalexin remain above the minimum inhibitory concentration (MIC) of MSSA. A range of MICs will be directly measured, with an expected range from 0.125 to 4.

SECONDARY OUTCOMES:
Clearance (CL/F) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the Clearance, or CL/F (L/h/kg), of both drugs.
Volume of Distribution (V/F) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the Volume of Distribution, or V/F (L/kg), of both drugs.
Half life (T1/2) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the half life, or T1/2 (hours), of both drugs.
Area under the curve (AUC) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the area under the curve, or AUC (h*mg/L), of both drugs.
Peak serum drug concentration (Cmax) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the peak serum drug concentration, or Cmax (mg/L), of both drugs.
Minimum serum drug concentration (Cmin) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the minimum serum drug concentration, or Cmin (mg/L), of both drugs.
Time at which maximal drug concentration is achieved (Tmax) of cefadroxil and cephalexin | Serum drug levels obtained at: 1, 2, 6, 8 hours (cephalexin); and 1, 2, 6, 8, 12 hours (cefadroxil)
  In defining pharmacokinetic parameters for both cephalexin and cefadroxil, the investigators will assess the time at which maximal drug concentration is achieved, or Tmax (hours), of both drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haynes, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No